CLINICAL TRIAL: NCT00003301
Title: A Dose Finding and Safety/Efficacy Trial of CPT-11 (Irinotecan) in Patients With Recurrent Malignant Gliomas
Brief Title: Irinotecan in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066241; NABTT-9711; JHOC-NABTT-9711
Record Dates: First submitted 1999-11-01; First posted 2004-04-09 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2005-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of irinotecan in treating patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of intravenous irinotecan when administered weekly for 4 weeks in patients with recurrent malignant gliomas. II. Describe the pharmacokinetics of this route of administration, measuring both irinotecan and the active metabolite SN-38, and determine the effects of hepatic enzyme inducing drugs, such as anticonvulsants, on the pharmacokinetics in these patients. III. Determine preliminary response data and activity of irinotecan in this patient population. IV. Correlate response with topoisomerase I levels in brain tumor tissue from patients undergoing treatment.

OUTLINE: Patients are stratified based on their use/kind of anticonvulsant drugs. This stratification yields two arms for this study. Arm I consists of patients who use anticonvulsant drugs that induce hepatic metabolic enzymes. Arm II consists of patients who use anticonvulsant drugs that cause modest to no induction of hepatic metabolic enzymes or no anticonvulsant drug. Three patients in each arm receive irinotecan by 90-minute IV infusions every week for 4 weeks, followed by a 2 week rest period. The dose is escalated for the next cohort of 3 patients in the absence of unacceptable dose limiting toxicity. The 6 week course is repeated until unacceptable toxicity or disease progression. Once the maximum tolerated dose has been established for each arm, additional patients are treated at that dose level. Patients are followed every 2 months.

PROJECTED ACCRUAL: A minimum of 3 patients will be accrued into the phase I portion of the study and a total of 18-35 patients will be accrued into each arm of the phase II portion of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant glioma that is progressive or recurrent following radiation therapy or chemotherapy Anaplastic astrocytoma Glioblastoma multiforme Low grade glioma that has progressed to biopsy proven high grade glioma is eligible if the progression occurred after radiotherapy with or without chemotherapy Measurable progression or recurrence by serial MR or CT imaging

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Greater than 2 months Hematopoietic: Absolute neutrophil count 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 4 times upper limit of normal Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: No uncontrolled hypertension No angina pectoris No evidence of uncontrolled cardiac dysrhythmia Other: No serious infection or other medical illness No other prior or concurrent malignancy within 5 years except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior topoisomerase 1 inhibitor (topotecan, irinotecan, 9- aminocamptothecin) No more that 1 prior chemotherapy regimen At least 6 weeks since nitrosourea and recovered At least 3 weeks since any other chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 3 months since completion of most recent course of radiotherapy and recovered Surgery: Not specified Other: No concurrent investigational agents At least 14 days since prior valproic acid No concurrent valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, MPH, Study Chair — Massachusetts General Hospital
Locations (9):
- United States (9):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Batchelor TT, Gilbert MR, Supko JG, Carson KA, Nabors LB, Grossman SA, Lesser GJ, Mikkelsen T, Phuphanich S; NABTT CNS Consortium. Phase 2 study of weekly irinotecan in adults with recurrent malignant glioma: final report of NABTT 97-11. Neuro Oncol. 2004 Jan;6(1):21-7. doi: 10.1215/s1152851703000218. PMID 14769136